CLINICAL TRIAL: NCT05318274
Title: Hypofractionated Radiation Therapy (1 Week) Compared With Standard Treatment (3.1 Weeks), Evaluation of Local Control of Breast Cancer Treated With Conservative Surgery.
Brief Title: Hypofractionated Radiation Therapy vs Standard Treatment in Breast Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Patricia Berenice Bolado Garcia, MD., Coordinación de Investigación en Salud, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2021-3203-005
Record Dates: First submitted 2022-02-23; First posted 2022-04-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Ductal Breast Carcinoma in Situ; Invasive Breast Cancer; Early-stage Breast Cancer; Stage 0 Breast Cancer; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ | interventions — Radiation Dose Hypofractionation; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (Experimental): Radiotherapy treatment with high hypofractionation, 26 Gy in 5 fractions to the whole breast.
  Interventions: Radiation: Hypofractionated radiotherapy
- ARM II (Active Comparator): Radiotherapy treatment with standard hypofractionation, 42.5 Gy in 16 fractions with simultaneous integrated increase of 5.5 Gy to the tumor bed in high-risk patients.
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Ultra hypofractionated 26 Gy in 5 fractions applied once with daily port film.
  Other Names: Adjuvant Radiation Therapy; External Beam Radiotherapy; 3D Conformal Radiation Therapy; Intensity Modulated Radiation Therapy; IMRT Fixed Gantry Radiation Therapy; Hypofractionated Whole Breast Irradiation; Quality of Life Questionnaire: EORTC QLQ-BR23

SUMMARY:
An explanatory study comparing complementary treatment to breast conservative surgery with radiation therapy DCIS, T1-T2 N0 M0 (AJCC v8) 1 week schedule vs 3.1 weeks standard schedule, in order to determine the equivalence of local tumor control, survival, acute and chronic toxicity. Shorter curse of radiation therapy may lead to similar local control of tumor cells and lower rates of toxicity than 3.1 standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the effectiveness of hypofractionated radiotherapy (1 week) with standard treatment (3.1 weeks) in the local control of breast cancer treated with conservative surgery.

SECONDARY OBJECTIVES:

I. Identify the histological lineage of the tumor.

II. Identify the degree of differentiation of tumor cells.

III. Identify the presence and type of receptors (estrogen, progesterone, HER-2NEU) through immunohistochemistry.

IV. Measure the frequency of progression or recurrence.

V. Identify the site of progression or recurrence.

VI. Measure the frequency of toxicity in both groups.

VII. Classify toxicity according to its severity.

VIII. Classify toxicity according to chronological presentation, acute, subacute, or chronic.

IX. Measure quality of life in both groups according to the European Organization for Research and Treatment Cancer scale, Breast Cancer-Specific Quality of Life Questionnaire, (EORTC, QLQ-BR23).

X. Measure quality of life in both groups according to the Eastern Collaborative Oncology Group (ECOG) performance scale.

XI. Measure 5-year survival.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: will receive radiotherapy treatment with high hypofractionation, 26 Gy in 5 fractions to the whole breast.

ARM II: will receive radiotherapy treatment with standard hypofractionation, 42.5 Gy in 16 fractions with simultaneous integrated increase of 5.5 Gy to the tumor bed in high-risk patients.

After completion of treatments, patients will be followed: 2 weeks after final fraction, 6 weeks after final fraction, every 4 months for the next 5 years

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by histopathological report of ductal carcinoma in situ (DCIS) or invasive breast carcinoma.
* Treated with breast-conserving surgery and stage pT1-2 pN0 M0.
* Over 18 years.
* Patients who sign informed consent for research study.

Exclusion Criteria:

* Positive nodes.
* Clinical or pathological stage T3-T4.
* History of previous irradiation.
* Postoperative positive margin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with ductal carcinoma in situ or early breast cancer.
Enrollment: 72 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Identify the progression timing. | 5 years
  Quantify the time to progression through follow up in both groups
Identify the recurrence timing. | 5 years
  Quantify the time to recurrence through follow up in both groups

SECONDARY OUTCOMES:
Identify the histological lineage of the tumor | 14 Months
  Carcinoma InSitu or Invasive Carcinoma;
  1. - Adenocarcinoma
  2. - Other
Identify the degree of differentiation of tumor cells | 14 months
  Histologic grade identification using Scarff-Bloom-Richardson (SBR) scale
  1. Grade 1: 3-5 points
  2. Grade 2: 6-7 points
  3. Grade 3: 8-9 points
Identify the presence and type of receptors (estrogen, progesterone, HER-2NEU) through immunohistochemistry | 14 months
  Number of participants with presence of Luminal A, B, HER-2NEU enriched or triple negative immunohistochemistry subtype.
  1. Luminal A: RE (+), RP >20%, Ki67 <20% y HER 2 NEU (-)
  2. Luminal B: RE (+), RP <20%, Ki67 >20% y HER 2 NEU (+/-)
  3. HER-2 Enriched: RE (-), RP (-),Ki67 any, HER 2 NEU (+)
  4. Triple Negative: RE (-), RP (-), Ki67 any, HER-2 (-)
Measure the frequency of toxicity in both groups. | 5 years
  Quantify the presence of toxicity categorized by CTCAE version 5 system.
  1. Grade 1: characterized by the presence of a mild adverse event that does not require treatment
  2. Grade 2: considers a moderate adverse event that may require medical treatment on an outpatient basis
  3. Grade 3: is a serious adverse event that should receive medical treatment, and even hospital treatment.
  4. Grade 4: is an adverse event with risk of death or disability that requires specialized medical management and hospitalization.
  5. Grade 5: considers the presence of death associated with an adverse event.
Classify toxicity according to its severity. | 5 years
  Quantify toxicity according to its severity categorized by CTCAE version 5 system.
  1. Dry skin: A disorder characterized by flaky and dull skin; the pores are generally fine, the texture is a papery thin texture
     - Grade 1 to 3
  2. Eczema: A disorder characterized by skin which becomes itchy, red, inflamed, crusty, thick, scaly, and/or forms blisters.
     - Grade 1 to 3
  3. Skin hyperpigmentation: A disorder characterized by darkening of the skin due to excessive melanin deposition.
     - Grade 1 to 2
  4. Dysphagia: A disorder characterized by difficulty in swallowing.
     - Grade 1 to 4
  5. Cough: A disorder characterized by sudden, often repetitive, spasmodic contraction of the thoracic cavity, resulting in violent release of air from the lungs and usually accompanied by a distinctive sound.
     - Grade 1 to 3
  6. Pneumonitis: A disorder characterized by inflammation focally or diffusely affecting the lung parenchyma.
     * Grade 1 to 5

OTHER OUTCOMES:
Breast Cancer-Specific Quality of Life Questionnaire, (EORTC, QLQ-BR23). | 5 Years
  Quantify quality of life with QLQ-BR23 questionnaire created by the European Organization for Research and Treatment of Cancer Group
Measure quality of life in both groups according to the European Organization for Research and Treatment Cancer scale (ECOG) | 5 Years
  Quantify quality of life with Eastern Cooperative Oncology Group (ECOG) Performance Status Scale

CONTACTS AND LOCATIONS:
Overall Officials: Fernando H Castillo-Lopez, Phy., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad Medica de Alta Especialidad, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No